CLINICAL TRIAL: NCT01453309
Title: Cost Effectiveness and Clinical Utility of Cell Saver Use for Two to Three Level Lumbar Fusions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Norton Leatherman Spine Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-N0216
Record Dates: First submitted 2011-10-10; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Low Back Pain Unresponsive to Non-surgical Care
Keywords: lumbar fusion; transfusion; cell-saver; cost-effectiveness
MeSH Terms: interventions — Operative Blood Salvage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cell Saver (Active Comparator): Patients will have the use of a cell-saver during surgery
  Interventions: Procedure: Cell Saver
- No Cell saver (Placebo Comparator): Patient will not have cell saver available during surgery.
  Interventions: Procedure: No Cell Saver

INTERVENTIONS:
Procedure: Cell Saver — Cell Savers are used intraoperatively to decrease the risk of transfusion due to surgical blood loss. Blood collected from the operative field is anticoagulated, filtered, and stored in a reservoir. Once a set volume of blood has been collected in the reservoir, the blood is separated into its red blood cell and plasma components by use of a centrifuge. Red blood cells are washed with a crystalloid solution and then reinfused into the patient.
  Arms: Cell Saver
Procedure: No Cell Saver — Cell Saver will not be available during surgery
  Arms: No Cell saver

SUMMARY:
The purpose of this study is to determine the cost-effectiveness of using a cell saver for 2 to 3 level lumbar fusions. A secondary objective is to determine if there will be a decrease in the number of allogenic blood transfusions when a cell saver is used intraoperatively. Another secondary objective is to determine incidence of complications associated with cell saver use and transfusions.

DETAILED DESCRIPTION:
INTRODUCTION:

Cell Savers are used intraoperatively to decrease the risk of transfusion due to surgical blood loss. Blood collected from the operative field is anticoagulated, filtered, and stored in a reservoir. Once a set volume of blood has been collected in the reservoir, the blood is separated into its red blood cell and plasma components by use of a centrifuge. Red blood cells are washed with a crystalloid solution and then reinfused into the patient. Although the theoretical benefits of using a cell saver are attractive, the literature seems to be controversial with respect to efficacy and cost-effectiveness. The benefits are clear in patients undergoing fusions for scoliosis that involve more than 5 levels where blood loss is considered substantial. It is less clear in patients who undergo a more limited two to three level lumbar fusion.

The purpose of this study is to determine the cost-effectiveness of using a cell saver for 2 to 3 level lumbar fusions. A secondary objective is to determine if there will be a decrease in the number of allogenic blood transfusions when a cell saver is used intraoperatively. Another secondary objective is to determine incidence of complications associated with cell saver use and transfusions.

METHODS Patients seen at the Norton Leatherman Spine Center scheduled to have decompression and fusion over 2 to 3 lumbar spine segments will be screened for the study. After obtaining informed consent, patients will be randomized to have a cell saver used intraoperatively (Cell Saver group) or no cell saver (Non-Cell Saver group). Data to be collected will include age, gender, smoking status, height, weight, co-morbidities, the use of medications that may increase bleeding (Plavix, Coumadin, Warfarin), or increase blood production (Ferrous sulfate, erythropoietin) medications used to decrease intraoperative bleeding (Aprotinin, Tranexamic Acid); the use of hypotensive anesthesia, ASA Grade, indications for surgery, date of surgery, estimated blood loss, surgical approach, surgical levels, bone graft used, operative time, complications, length of stay, discharge information, whether or not patient pre-donated blood, hemoglobin, hematocrit and maximum body temperature prior to surgery and during the patient's hospital stay, surgical drain output, products transfused intraoperatively and postoperatively and the amount of cell saver salvaged, re-infused, and the cell-saver hematocrit and hemoglobin prior to re-infusion. The costs associated with the use of the cell-saver and/or blood transfusions, including supplies and personnel time, will be determined.

Randomization Randomization will be through stratified block randomization to allow for stratification of the number of levels fused. Randomization will use sealed envelopes.

Sample Size To detect a medium effect size of 0.3 with an α error of 0.05, a total of 220 subjects need to be included in the analysis. To account for subject withdrawal, a total of 240 subjects will be enrolled

Procedures Patients receiving care at the Norton Leatherman Spine Center will be screened as potential subjects for the study. Only the existing information obtained per standard routine medical procedures will be used. Patients who fail pre-screening will not be recorded on any log or form. Patients considered potential candidates for the study based on screening will sign an Institutional Review Board -approved Informed Consent Document and HIPAA Authorization form prior to participating in any study activity.

Subjects will be randomized to receive or not receive cell saver during surgery. The following data will be collected during the clinic visit: age, gender, smoking status, height, weight, co-morbidities, the use of medications that may increase bleeding (Plavix, Coumadin, Warfarin), or increase blood production (Ferrous sulfate, erythropoietin). The following pre-operative data will be collected: hemoglobin, hematocrit, body temperature and whether or not patient pre-donated blood, the predonated blood volume and date of donation.

Surgery will be performed per the standard of care of the treating surgeon. The choice of surgical approach, instrumentation and bone grafts/bone graft substitutes will be at the discretion of the surgeon. The following intraoperative data will be collected: use of hypotensive anesthesia, ASA Grade, indications for surgery, date of surgery, estimated blood loss, surgical approach, surgical levels, bone graft used, operative time products transfused intraoperatively. In the subjects randomized to the Cell Saver group, the amount of cell saver salvaged, re-infused, and the cell-saver hematocrit and hemoglobin prior to re-infusion will be determined and collected. In-hospital post-operative data to be collected include: complications, length of stay, discharge information, hematocrit, hemoglobin and maximum body temperature during the patient's hospital stay, surgical drain output, products transfused postoperatively.

Subjects will be transfused at a set transfusion threshold of hemoglobin of 7.0g/dL or below and corresponding hematocrit of 21 or below. Subjects with Hb 7.0g/dL and are symptomatic as evidenced by tachycardia, hypotension, orthostatic hypotension or have pre-existing cardiac or pulmonary disease will also be transfused.

The risks that occur in this study are associated with the general risks of spine surgery. Risks associated with allogeneic blood transfusion include allergic reactions, hemolytic reactions, isoimmunization, graft versus host reactions, increased infection rates, and transmission of bloodborne pathogens, including human immunodeficiency virus and hepatitis. Risks associated with the use of a cell saver include a paradoxical increase in blood loss, electrolyte depletion, metabolic acidosis, and hematuria

Endpoints The primary endpoint is the volume of blood transfusion required. Secondary endpoints include

* Immediate post-op Hematocrit level
* Immediate post-op Hemoglobin level
* Volume of blood products used post-operatively

Statistical Analysis Descriptive statistics, including frequency counts for discrete variables and measures of central tendency (means, medians) and dispersion (standard deviation, range) for continuous variables will be calculated. Comparisons between the Cell Saver and non-Cell Saver groups will be done with independent t test for continuous variables and χ2 tests for discrete variables. To determine the effects of potentially confounding variables, analysis of covariance to compare the Cell Saver and non-Cell Saver groups will be used. This will help identify variables that may be statistically different between the Cell Saver and non-Cell Saver groups that could potentially influence the total units of blood transfused. Those variables that were significantly related (i.e., correlated) with the number of units of blood transfused will be entered as covariates into the statistical model to determine if they affect the statistical conclusions between the Cell Saver and non-Cell Saver groups. All analyses will performed an a priori alpha level of 0.05 using IBM SPSS version 19.0.

Funding This study will be unfunded.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at time of enrollment
* Signed informed consent
* Requires fusion of 2 to 3 levels from L1-S1 for degenerative lumbar disorders

Exclusion Criteria:

* Spinal trauma/fracture/malignancy
* Infection as an indication for surgery
* Pregnant or nursing women
* Prisoners
* Institutionalized in a non-voluntary and/or dependent residence (including hospitals, group homes, etc.), who may not be competent to give informed consent.
* Inability to speak or understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Volume of blood transfused | Hospitalization, range of 3 to 14 days
  The total volume of blood and blood products transfused during surgery an during hospitalization will be determined

SECONDARY OUTCOMES:
Immediate post-op Hematocrit level | Post-operative, range of 1 to 14 days
  Immediate post-op Hematocrit level
Immediate post-op Hemoglobin level | Post-operative, range of 1 to 14 days
  Immediate post-op Hemoglobin level

CONTACTS AND LOCATIONS:
Overall Officials: Mladen Djurasovic, MD, Principal Investigator — Norton Leatherman Spine Center
Locations (1):
- Norton Leatherman Spine Center, Louisville, Kentucky, United States